CLINICAL TRIAL: NCT06027840
Title: A Preliminary Test of Concurrent vs. Sequential Cessation of Dual Cigarette and E-cigarette Use on Behavior, Tobacco Toxicant Exposure, and Health Effects
Brief Title: Concurrent vs. Sequential Cessation of Dual Cigarette and E-cigarette Use
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000035713; 2P50CA196530-06 (NIH)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cigarette Smoking; E-Cigarette Use; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Vaping; Smoking Cessation | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QUIT-C (Concurrent) (Experimental): Treatment in this arm will emphasize concurrent cessation of cigarettes and e-cigarettes. All participants will receive 12-weeks of varenicline, weekly individual counseling, and access to cessation resources including a guided self-change booklet and links to free text-based support. Counseling and cessation resources will emphasize concurrent cessation.
  Interventions: Drug: Varenicline; Behavioral: Counseling; Behavioral: Guided Self-Change Booklets
- QUIT-S (Sequential) (Experimental): Treatment in this arm will focus on cessation of cigarettes followed sequentially by cessation of e-cigarettes. All participants will receive 12-weeks of varenicline, weekly individual counseling, and access to cessation resources including a guided self-change booklet and links to free text-based support. Counseling and cessation resources will emphasize sequential cessation.
  Interventions: Drug: Varenicline; Behavioral: Counseling; Behavioral: Guided Self-Change Booklets

INTERVENTIONS:
Drug: Varenicline — Varenicline prescription will follow the standard induction period: varenicline 0.5 mg once per day for Days 1-3, varenicline 0.5 mg twice per day for Days 4-7, then varenicline 1 mg twice per day (when varenicline reaches peak efficacy for tobacco cessation). Participants will remain on varenicline for 12 weeks total. Dose adjustments (e.g., reduction to 0.5 mg twice per day if 1 mg is not well tolerated) will be allowed at the discretion of the clinical pharmacist/APRN/physician.
Behavioral: Counseling — Tobacco Treatment Service clinicians will deliver weekly counseling sessions, monitor participants for adverse events, and record participants' weekly cigarette and e-cigarette use. At the first counseling session clinicians will review medication proper use instructions, and potential side effects and strategies to address them at the first counseling session. Study medication refills will be distributed at 4-week intervals. Sessions will focus on quit plan preparation, supportive and practical cessation counseling, resetting quit dates, and relapse prevention.
Behavioral: Guided Self-Change Booklets — The booklet includes information on how to reduce and quit both cigarettes and e-cigarettes on their own, how to prevent relapse, how to set a quit date, and how to enroll in text-based support resources.

SUMMARY:
The purpose of this research study is to understand whether concurrent treatment for cigarettes and e-cigarettes in which an individual quits both products at the same time (QUIT-C) or sequential treatment in which an individual quits cigarettes first followed by e-cigarettes is more effective for quitting both products. The study will also compare the effect of treatment on health-related biomarkers. All participants will receive varenicline, a medication used to treat tobacco use dependence, counseling, and cessation resources (i.e., links to text-based support, self-change booklet). Varenicline helps to reduce cravings for tobacco use and decreases the pleasurable effects of cigarettes and other tobacco products.

DETAILED DESCRIPTION:
Inclusion/exclusion criteria will be determined via initial online screening and then confirmed with tele-video/phone call final screening. Non-pregnancy verification will be ascertained via remote pregnancy test.

All participants will be asked to provide assessments (as described below) throughout the sampling process to assess cigarette smoking and e-cigarette use behavior, varenicline use, and use of cessation resources.

This is a 12 week, open-label study of varenicline.

ELIGIBILITY:
Inclusion Criteria:

* English literate
* Report cigarette smoking, and e-cigarette use for at least the past 3 months
* Smoke 5 or more cigarettes per day
* Report e-cigarette use for at least 14 days in the past month
* Interested in quitting both products in the next month and willing to set a quit date.

Exclusion Criteria:

* Vulnerable Populations: Investigators will not be enrolling vulnerable populations, specifically pregnant women, children, prisoners, or institutionalized individuals
* Investigators also will not enroll participants incapable of providing their own consent. The rationale will be provided to the individual as well as his or her family members. Referrals for further evaluation, including urgent or emergent evaluation, will be made as needed and clinically warranted.
* Investigators will exclude anyone currently using any smoking cessation services and/or FDA pharmacotherapies.
* Verification of Non-Pregnancy: Females ages <55 will be given a commercially available pregnancy test to verify non-pregnancy. A female of child-bearing age that is currently pregnant or breastfeeding or report an unwillingness to use effective birth control (i.e., abstinence, IUD, implant, sterilization, pill, patch, ring, or barrier method such as condoms with spermicide) for the duration of the study will not be enrolled.
* Individuals using other tobacco or nicotine products besides cigarettes and e-cigarettes > once per week in the last 30 days will be excluded.
* Investigators will exclude individuals with medical contraindications for varenicline use (i.e., severe renal impairment and unstable cardiac history)
* Medical Conditions: Investigators will not enroll anyone with a current, serious uncontrolled medical/psychiatric condition (e.g., a condition that required a hospitalization or intensive outpatient treatment in the past year) based on review by Study Physician that would increase risk of severe adverse events and/or interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cigarette Abstinence at Week 12- Carbon Monoxide | Week 12
  7-day point prevalence cigarette abstinence at Week 12, biochemically verified by breath carbon monoxide

SECONDARY OUTCOMES:
E-Cigarette Abstinence at Week 12- Cotinine | Week 12
  7-day point prevalence e-cigarette abstinence at Week 12, biochemically verified by urine cotinine
Number of cigarettes smoked per day | Baseline up to week 12
  Number of cigarettes smoked per day assessed by self-report
Percent days of e-cigarette usage | Baseline up to week 12
  Percent days of e-cigarette usage assessed by self-report
Biomarkers of tobacco-related harm exposure | Baseline up to week 12
  Primary urinary biomarkers of tobacco-related harm exposure will be assessed including NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol), a tobacco carcinogen linked to lung cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No